CLINICAL TRIAL: NCT03345771
Title: Antimicrobial Barrier Dressing Versus Closed-incision Negative Pressure Therapy in the Obese Primary Total Joint Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00496
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antimicrobial Barrier Dressing (Active Comparator): postoperative wound dressing with either anti-microbial dressing placed in the operating room from surgery to postoperative day 7
  Interventions: Combination Product: Antimicrobial Barrier Dressing
- Closed-incision Negative Pressure Therapy (Active Comparator): portable NPWT device placed in the operating room from surgery to postoperative day 7
  Interventions: Device: Negative Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Combination Product: Antimicrobial Barrier Dressing — Ionic Silver is a soft, nonwoven pad or ribbon that features the gelling benefits of Hydrofiber technology plus antimicrobial ionic silver.
  Other Names: AQUACEL Ag Hydrofiber Dressing
  Arms: Antimicrobial Barrier Dressing
Device: Negative Pressure Wound Therapy (NPWT) — PICO provides suction known as negative Pressure wound Therapy (NPWT) which draws out excess fluid from a wound and protects the injured area from getting dirty to ultimately help promote healing. PICO consists of an nPwT pump connected to an absorbent gentle adhesive dressing
  Other Names: PICO
  Arms: Closed-incision Negative Pressure Therapy

SUMMARY:
The purpose of this study is to determine whether an occlusive antimicrobial barrier dressing or portable negative pressure wound dressing is superior in preventing wound complications and infection rates in obese patients undergoing total joint arthroplasty (TJA). Approximately 240 subjects (120 for total knee arthroplasty and 120 for total hip arthroplasty) will be enrolled to evaluate the outcomes associated with silver impregnated dressings and negative pressure wound therapy (NPWT) in treating this subset of patients and analyze the cost benefit of each.

ELIGIBILITY:
Inclusion Criteria:

* Those identified at pre-operative testing to have an elevated BMI (> 35)

Exclusion Criteria:

* Active infection
* previous scar or wound healing complication
* post traumatic degenerative joint disease (DJD) with hardware
* revision surgery
* inflammatory arthritis
* anticoagulation outside of the standard of care.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antimicrobial Barrier Dressing | Closed-incision Negative Pressure Therapy
Started | 115 | 115
Completed | 115 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antimicrobial Barrier Dressing | Closed-incision Negative Pressure Therapy | Total
Number analyzed (Participants) | 115 | 115 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.87 (9.84) | 60.87 (9.32) | 60.24 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 82 | 82 | 164
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 115 | 115 | 230
Region of Enrollment [Number; unit: participants]
  United States | 115 | 115 | 230

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Score
Description: A patient is asked to indicate his/her perceived scar severity along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (worst possible scar) to 100 (best possible scar); the higher the score, the better the scarring.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antimicrobial Barrier Dressing | Closed-incision Negative Pressure Therapy
Number analyzed (Participants) | 78 | 81
score on a scale | 64 (26) | 61 (24)

2. Primary Outcome: Wound Evaluation Scale (WES)
Description: WES is a 6-item scale. Items 1-5 are scored 0 (yes) or 1 (no), and item 6 is scored 0 (poor) or 1 (acceptable). The total score range is 0-6; the higher the score, the more optimal the wound healing.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antimicrobial Barrier Dressing | Closed-incision Negative Pressure Therapy
Number analyzed (Participants) | 50 | 42
score on a scale | 4.3 (1.3) | 4.2 (1.7)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Study members will monitor the participants for adverse events on an ongoing basis
Arm/Group | Antimicrobial Barrier Dressing | Closed-incision Negative Pressure Therapy
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/115
Serious Adverse Events (participants affected / at risk) | 3/115 | 0/115
Other Adverse Events (participants affected / at risk) | 6/115 | 2/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antimicrobial Barrier Dressing (N=115) | Closed-incision Negative Pressure Therapy (N=115)
Irrigation and Debridement (Surgical and medical procedures) | 2 | 0
Revision Total Knee Arthroplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antimicrobial Barrier Dressing (N=115) | Closed-incision Negative Pressure Therapy (N=115)
Wound drainage (Surgical and medical procedures) | 5 | 2
Non-healing wound (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03345771/Prot_SAP_000.pdf